CLINICAL TRIAL: NCT05220020
Title: Prospective, Randomized Controlled, Single-center, Phase III Clinical Study of TACE Combined With Lenvatinib Versus TACE Sequential Lenvatinib in the Treatment of Intermediate/Advanced Liver Cancer
Brief Title: TACE Combined With Lenvatinib Versus TACE Sequential Lenvatinib in the Treatment of Intermediate/Advanced Liver Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Zhao, Associate Director of Minimally Invasive Intervention, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2021-370-01
Record Dates: First submitted 2022-01-12; First posted 2022-02-02 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: TACE; Lenvatinib; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Synchronous treatment group: the first course of TACE treatment was started after 2-3 weeks Lenvatinib treatment.
  Interventions: Procedure: TACE(Transcatheter arterial chemoembolization); Drug: Lenvatinib
- Control group (Active Comparator): Sequential treatment group: patients with uncontrolled TACE progression after TACE treatment were sequentially treated with Lenvatinib.
  Interventions: Procedure: TACE(Transcatheter arterial chemoembolization); Drug: Lenvatinib

INTERVENTIONS:
Procedure: TACE(Transcatheter arterial chemoembolization) — Hepatic arterial chemoembolization treatment
Drug: Lenvatinib — Experimental group(Synchronous treatment group): the first course of TACE treatment was started after 2-3 weeks Lenvatinib treatment.Control group:(Sequential treatment group)patients with uncontrolled TACE progression after TACE treatment were sequentially treated with Lenvatinib.
  Other Names: Lenvatinib oral

SUMMARY:
TACE(transcatheter arterial chemoembolization) has been recommended by domestic and international guidelines as the standard treatment for a subset of HCC patients with very high heterogeneity, including BCLC stage B(intermediate-stage) and some BCLC stage C(advanced-stage). However, for these patients, TACE therapy alone is often difficult to achieve satisfactory efficacy. Moreover, in the course of repeated TACE treatment, tumor remission rate continues to decrease, and drug resistance and liver function damage are prone to be aggravated.Studies have shown that TACE and TKI combined therapy can not only inhibit the release of VEGF and other angiogenic growth factors after TACE, but also prolong the interval of TACE treatment、reduce the frequency of TACE treatment by inhibiting residual tumor proliferation, thus reducing liver function damage.Lenvatinib therapy,which is associated with a high response rate compared with Sorafinib and the cost-effect advantage of Lenvatinib was significantly better than that of sorafenib.But it has not been determined whether lenvatinib should be used synchronously or sequentially based on TACE.Through the comparative study of different timing combinations, we explore the interventional timing of Lenvatinib in intermediate-advanced liver cancer, providing a new scheme for interventional combination therapy.

DETAILED DESCRIPTION:
Femoral artery puncture and catheterization were performed in every cycle of treatment,a catheter was inserted and located in feeding hepatic artery of tumor. The therapeutic scheme was that, synchronous treatment group(experimental group): the first course of TACE treatment was started after 2-3 weeks Lenvatinib treatment.Sequential treatment group(control group): patients with uncontrolled TACE progression after TACE treatment were sequentially treated with Lenvatinib.TACE was repeated on demand and continued until disease progression or unacceptable toxicity.Follow-up was performed every 3 months after disease stabilization until disease progression. When tumor progression occurs, subjects should follow the second-line or third-line regimen recommended in the current clinical guidelines for the diagnosis and treatment of liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent form (ICF) and any locally required authorization obtained from the patient prior to any mandatory study specific procedures, sampling, and analyses.
* Provision of signed and dated written genetic informed consent prior to optional collection of sample for genetic analysis.
* Patients with BCLC stage C hepatocellular carcinoma confirmed by pathology or clinically diagnosed
* Anticipated life expectancy ≥ 12 months
* Eligible for TACE treatment, including BCLC-B, and BCLC-C only for Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* No prior systemic therapy (including systemic investigational agents) for HCC, especially immunotherapy
* Age ≥18 years and < 75 years at the time of screening.
* Portal vein invasion or extrahepatic oligosaccharides were detected by baseline imaging. Oligosaccharides were defined as no more than two extrahepatic organs and no more than three tumors.
* Portal vein thrombosis visible on baseline/eligibility imaging, patients with Vp1 and Vp2 are included
* Patients who have previously undergone surgical resection, thermal ablation and other radical therapies for liver cancer may be enrolled. Prior TACE therapy must be used as part of the radical therapy (e.g. in combination with thermal ablation or surgery), but not as the sole form of previous treatment. These treatments need to be completed one month before enrollment.
* Child-Pugh score class A to B7
* No local antitumor therapy for hepatocellular carcinoma was received within 4 weeks prior to enrollment
* No evidence of extrahepatic disease on any available imaging
* No previous systemic antitumor therapy for hepatocellular carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment
* The expected survival time is no less than 3 months
* BCLC Stage B: Patients with Intermediate HCC exceeding the "up-to-seven" criteria [i.e., the sum of tumor number (number) and maximum tumor diameter (cm) exceeds 7]
* Patients with HBV infection, which is characterized by positive hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibodies (anti-HBcAb) with detectable HBV DNA (≥10 IU/ml or above the limit of detection per local lab standard), must be treated with antiviral therapy, as per institutional practice. HBV antiviral therapy must be initiated prior to randomization and patients must remain on antiviral therapy for the study duration and for 6 months after the last dose of study medication. Patients must show evidence HBV stabilization or signs of viral response (e.g., reduction HBV DNA levels) prior to starting IP. Patients who test positive for anti-hepatitis B core (HBc) with undetectable HBV DNA (<10 IU/ml or under the limit of detection per local lab standard) do not require anti-viral therapy prior to randomization. These subjects will be tested at every cycle to monitor HBV DNA levels and initiate antiviral therapy if HBV DNA is detected (≥10 IU/ml or above the limit of detection per local lab standard). HBV DNA detectable subjects must initiate and remain on antiviral therapy for the study duration and for 6 months after the last dose of study medication.
* Patients with HCV infection must have management of this disease per local institutional practice throughout the study. HCV diagnosis is characterized by the presence of detectable HCV ribonucleic acid (RNA) or anti-HCV antibody upon enrollment.
* At least 1 measurable intrahepatic lesion suitable for repeat assessments according to the following mRECIST criteria: （1）Liver lesions that show typical features of HCC on IV contrast-enhanced CT or MRI scans, ie, hypervascularity in the arterial phase with washout in the portal or the late venous phase；（2）Viable, non-necrotic portion (arterial phase IV contrast-enhancing) that can be accurately measured at baseline as ≥10 mm in the longest diameter.
* Adequate organ and marrow function as defined below. Criteria "a," "b," "c," and "f" may not be met with transfusions, infusions, or growth factor support administered within 14 days of starting the first dose.

Hemoglobin ≥9.0 g/dL、Absolute neutrophil count ≥1000/µL、Platelet count ≥50000/µL、Total bilirubin ≤2.0 × the upper limit of normal (ULN)、alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5 × ULN、Albumin ≥2.8 g/dL、International normalized ratio ≤1.6、2+ proteinuria or less urine dipstick reading、Calculated creatinine clearance (CL) ≥30 mL/min as determined by Cockcroft-Gault (using actual body weight) or 24hour urine creatinine CL

Males:

Creatinine CL = Weight (kg) × (140 - Age) (mL/min) 72 × serum creatinine (mg/dL)

Females:

Creatinine CL = Weight (kg) × (140 - Age) × 0.85 (mL/min) 72 × serum creatinine (mg/dL)

* Must have a life expectancy of at least 12 weeks.
* Body weight >30 kg

Exclusion Criteria:

* Evidence of macrovascular invasion (MVI).
* Evidence of extrahepatic spread (EHS)
* Being a candidate for curative treatments (e.g. surgical resection, RFA or liver transplantation).
* Any condition representing a contraindication to TACE as determined by the investigators(for example, the main portal vein obstruction without collateral vessels formed, etc.);
* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC;History of leptomeningeal disease;
* Allergy to TACE process medications (such as contrast agents) or to Lenvatinib is known or suspected
* There are obvious arteriovenous fistula or portal vein fistula in the liver.
* Tumor invasion or oppression of the common bile duct, resulting in malignant obstructive jaundice;
* Tumor volume of 70% or more of the liver;
* Previous history of molecular targeted therapy, such as sorafenib, apatinib, etc.
* Patients who had previously used systemic therapy (e.g., immunotherapy, targeted therapy) were excluded from the study
* Severe heart conditions, such as congestive heart failure & GT; New York Heart Association (NYHA) Class II, active coronary artery disease (patients with myocardial infarction that occurred 6 months prior to enrollment), arrhythmias requiring treatment (other than beta-blockers, calcium antagonists, or digoxin); Uncontrolled hypertension (diastolic blood pressure not below 90mmHg even after treatment with 3 antihypertensive drugs;
* Active clinical severe infection (> Level 2 NCI-CTCAE version 4.0);
* Presence of active pulmonary tuberculosis or inability to exclude intrapulmonary lesions of old pulmonary tuberculosis.
* Known tumors of the central nervous system, including brain metastases;
* Clinically significant gastrointestinal bleeding within 30 days prior to enrollment;
* Autoimmune disease (HIV);
* Pregnant or breast-feeding patients;
* Prior history of liver transplantation;
* Any unstable condition or condition that may compromise the patient's safety and his/her compliance with the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Two-Years Overall Survival Rate | Two-Years
  Percentage of patients who survived two years after inclusion

SECONDARY OUTCOMES:
Two-years progression-free survival rate | Two-years
  It is defined as the percentage of patients who achieve a time interval of two years of no disease progression (i.e., intrahepatic recurrence or extrahepatic metastasis) or death (by any cause) from date of enrollment, whichever occurs first.
Objective response rate | Two-years
  The percentage of patients who achieved a complete or partial response at some point in their life
Evaluate the patients cancer-related QoL using the European Organization for Research and Treatment of Cancer (EORTC) QOL questionnaire (QLQ), the EORTC QLQ-HCC18. | From date of randomization up to two years, approximately
  Change in sub-scale and total scores of EORTC QLQ-HCC18 from baseline through follow-up.
Progressive survival to TACE intolerance(TTUP，time to TACE-untreatable progression) | From date of randomization up to two years, approximately
  From randomization to the time when the patient first developed child-Pugh grade C liver function for any reason, ECOG score exceeding 2, portal main vein or vena cava cancer thrombus formation, and extrahepatic metastasis
Evaluate the patients cancer-related QoL using the European Organization for Research and Treatment of Cancer (EORTC) QOL questionnaire (QLQ), the EORTC QLQ-C30. | From date of randomization up to two years, approximately
  Change in sub-scale and total scores of EORTC QLQ-C30 from baseline through follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhao, M.D. & Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Minimally Invasive and Interventional Radiology, Liver Cancer Study and Service Group, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China